CLINICAL TRIAL: NCT03608995
Title: Combined Detection of Interleukin-6 and Insulin-like Growth Factor Binding Protein-1 Total and Native (Premaquick) for the Prediction of Delivery in Women With Threatened Preterm Labor
Brief Title: Diagnostic Tests in the Context of Threatened Preterm Labour
Acronym: PREMAQUICK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Mr. Thierry PAPER - Biosynex Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CHU-394; 2018-A00619-46 (Other: 2018-A00619-46)
Record Dates: First submitted 2018-06-15; First posted 2018-08-01 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Preterm Labor; Immunochromatographic Assay; Predictive Value of Tests; Preterm Delivery; Biomarkers
Keywords: preterm labor; biomarkers; Preterm delivery threat
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Premaquick© (Experimental)
  Interventions: Diagnostic Test: Premaquick (Diagnostic test)
- Quikcheck (Other)
  Interventions: Diagnostic Test: Quikcheck fFN ™

INTERVENTIONS:
Diagnostic Test: Premaquick (Diagnostic test) — PREMAQUICK® is a rapid multiparametric test which aim to detect the presence of IGFBP-1 (Insulin-like Growth Factor-Binding Protein 1), fragmented IGFBP-1 and IL-6 (Interleukin 6) in vaginal secretions. By combining biomarkers of myometrial activation, cervical maturity and inflammation / infection, PREMAQUICK® integrates the main pathogenic mechanisms responsible for premature delivery, which makes it possible to predict or, on the contrary, rule out the risk of childbirth within 7 to 14 days. This test is intended for in vitro diagnostic use.
  Vaginal secretions are collected under speculum with a swab (10 seconds of impregnation of the swab). The swab is immersed in a tube containing an extraction buffer for 10 seconds. The tube is mixed and then 3 drops are deposited in each wells of the test device for 10 minutes. Visual reading should be done between 10 and 15 minutes.
  Arms: Premaquick©
Diagnostic Test: Quikcheck fFN ™ — - The Hologic QuikCheck fFN test is intended to be used for the qualitative detection of fetal fibronectin in cervicovaginal secretions. The presence of fetal fibronectin in cervicovaginal secretions between 22 weeks, 0 days and 34 weeks, 6 days of gestation is associated with elevated risk of preterm delivery. Quick Check fFN test® is a 10 min, one-step, visual test consists of a sterile polyester-tipped applicator, fetal fibronectin test strip, and sample extraction buffer. The QuikCheck fFN is a solid-phase immunogold assay which aim to detect fetal fibronectin. A positive specimen will result in two visible lines and a negative specimen will result in one visible line (control).
  Arms: Quikcheck

SUMMARY:
The primary purpose of the protocol is to compare the diagnostic accuracy in terms of positive and negative predictive values of Premaquick © (combined detection of IL-6 / IGFBP-1 total / IGFBP-1 native) and Quikcheck fFN ™ (fibronectin detection) tests for prediction of spontaneous delivery within 7 days in women with threatened preterm labor. The study hypothesis is that combined detection of IL-6 / IGFBP-1 total / IGFBP-1 native dice the admission will improve the prediction of delivery compared to the detection of fetal fibronectin alone in women with threatened preterm labor.

DETAILED DESCRIPTION:
The threat of premature labour is the main cause of hospitalization during pregnancy (38% of hospitalizations). To date, the assessment of severity relies mainly on ultrasound measurement of the cervix. The length of the cervix is significantly correlated with the risk of spontaneous premature delivery. A threshold of 25mm is relevant to rule out a delivery within 7 days but the identification of new markers including biological would be interesting to guide the clinician in assessing the risk of preterm birth. Among the biomarkers measured in vaginal secretions, the detection of fetal fibronectin seems to be the most relevant because of a high negative predictive value (NPV) up to 100% to rule out a delivery within 7 days. However, the use of this test is discussed because of its low positive predictive value (PPV) to predict delivery within 7 days (from 11% to 48%). The use of Premaquick © test (Biosynex, Strasbourg, France), which allow the simultaneous quantification of IL-6, total IGFBP-1 and native IGFBP-1 could be more efficient compared to the detection of fibronectin by improving the VPP. The results already obtained on a cohort of 97 patients (Eleje et al., 2016) show a similar NPV and a higher PPV of the Premaquick© test compared to the Quikcheck fFN ™ test (PPV up to 95% when the 3 markers are positive). Investigator wish to conduct a comparative study between these two tests on a larger cohort of patients (n = 220). Results of the tests will be masked for the clinician and the patient in order to assess and compare their ability to predict delivery within 7 days without modify the current medical management.

ELIGIBILITY:
Inclusion Criteria:

* Major pregnant women admitted to Clermont-Ferrand CHU maternity for threatened preterm delivery with intact membranes between 24 and 34 (+6 days) week of amenorrhea, with length of cervix < 30mm (ultrasound measurement).
* Ability to give informed consent.
* French social security scheme.

Exclusion Criteria:

* - Dilation of the cervix ≥ 4 cm
* Triple pregnancy or more
* Fetal membranes rupture
* Known uterine malformation
* Hydramnios
* Fetal malformation
* Placenta previa
* Abundant metrorrhagia
* Patient who had already participated in the study during the same pregnancy
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of Premaquick and Quikcheck fFN ™ tests to predict delivery within 7 days (yes / no). | Results of the tests are given by the biochemistry department after a minimum of 15 days after the tests have been performed. The date of delivery is obtained by analyzing the patient file.
  The results (positive / negative) of the Premaquick and Quikcheck fFN ™ tests and the delay between the test and delivery time (in days) will allow to determine the PPV and NPV of the tests to predict delivery within 7 days.

SECONDARY OUTCOMES:
Number of positive markers of the Premaquick test | up to 17 weeks
  Number of positive / negative markers (0, 1, 2 or 3)
Number of negative markers of the Premaquick test | up to 17 weeks
  Number of positive / negative markers (0, 1, 2 or 3)

CONTACTS AND LOCATIONS:
Overall Officials: Denis GALLOT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Compan C, Rossi A, Piquier-Perret G, Delabaere A, Vendittelli F, Lemery D, Gallot D. [Prediction of spontaneous preterm birth in symptomatic patients: A review]. J Gynecol Obstet Biol Reprod (Paris). 2015 Oct;44(8):740-51. doi: 10.1016/j.jgyn.2015.06.008. Epub 2015 Jun 29. French. PMID 26139036
- [Background] Deplagne C, Maurice-Tison S, Coatleven F, Vandenbossche F, Horovitz J. [Sequential use of cervical length measurement before fetal fibronectin detection to predict spontaneous preterm delivery in women with preterm labor]. J Gynecol Obstet Biol Reprod (Paris). 2010 Nov;39(7):575-83. doi: 10.1016/j.jgyn.2010.08.001. Epub 2010 Sep 29. French. PMID 20884131
- [Background] Eleje GU, Ezugwu EC, Eke AC, Eleje LI, Ikechebelu JI, Ezebialu IU, Obiora CC, Nwosu BO, Ezeama CO, Udigwe GO, Okafor CI, Ezugwu FO. Accuracy of a combined insulin-like growth factor-binding protein-1/interleukin-6 test (Premaquick) in predicting delivery in women with threatened preterm labor. J Perinat Med. 2017 Nov 27;45(8):915-924. doi: 10.1515/jpm-2016-0339. PMID 28236632
- [Background] Sentilhes L, Senat MV, Ancel PY, Azria E, Benoist G, Blanc J, Brabant G, Bretelle F, Brun S, Doret M, Ducroux-Schouwey C, Evrard A, Kayem G, Maisonneuve E, Marcellin L, Marret S, Mottet N, Paysant S, Riethmuller D, Rozenberg P, Schmitz T, Torchin H, Langer B. [Prevention of spontaneous preterm birth (excluding preterm premature rupture of membranes): Guidelines for clinical practice - Text of the Guidelines (short text)]. J Gynecol Obstet Biol Reprod (Paris). 2016 Dec;45(10):1446-1456. doi: 10.1016/j.jgyn.2016.09.011. Epub 2016 Nov 9. French. PMID 27836377